CLINICAL TRIAL: NCT06355388
Title: TRAnscutaneous vaGUS Nerve Stimulation in Patients With Chronic Heart Failure
Acronym: TRAGUS-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Toscana Gabriele Monasterio (Other)
Collaborators: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Michele Emdin, Professor, Fondazione Toscana Gabriele Monasterio
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TRAGUSHF
Record Dates: First submitted 2024-02-04; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure With Midrange Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In order to maintain the 'double-blind,' at the end of the experimental protocol, the data acquired in each phase (baseline, active tVNS, placebo tVNS) will be saved in three different files, made unrecognizable by one of the investigators not involved in the tabulation and data analysis. A second investigator, unaware of the stimulation phases, will proceed with the tabulation of the data for each individual recording (three per patient). Only at the end of the study (or after recruiting 50% of patients for any interim analyses), will the investigators responsible for data analysis be revealed the corresponding phase for each recording.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tVNS (Experimental): The ear clip of the device will be positioned at the level of the patient's tragus delivering current.
  Interventions: Device: Active tVNS
- Sham tVNS (Placebo Comparator): The ear clip of the device will be positioned at the level of the patient's tragus but not delivering current.
  Interventions: Device: Sham tVNS

INTERVENTIONS:
Device: Active tVNS — As for the short-term phase, the ear clip of the "Parasym" device (Parasym, London, United Kingdom), containing the stimulation electrode, will be positioned at the level of the patient's tragus, and a 10-minute stimulation will be initiated with a pulse width of 200 μs, a frequency of 30 Hz, and an intensity of one mA lower than the patient's sensitivity threshold.
  As fort he mid-term phase, a device will be given to the patient, which will be instructed to position the ear clip of the device at the level of the tragus and to set stimulation parameters as established in the laboratory (see above). Each patient will be asked to undergo at least one hour daily stimulation for a period of 4 weeks, reporting on a diary the timing and details of the each session.
  Arms: Active tVNS
Device: Sham tVNS — As for the short-term phase, the ear clip of the "Parasym" device (Parasym, London, United Kingdom), containing the stimulation electrode, will be positioned at the level of the patient's tragus for 10-minute but no current will be delivered.
  As fort he mid-term phase, a device (configured to withhold power delivery) will be given to the patient, which will be instructed to position the ear clip of the device at the level of the tragus and to set stimulation parameters as established in the laboratory (see above). Each patient will be asked to undergo at least one hour daily stimulation for a period of 4 weeks, reporting on a diary the timing and details of the each session.
  Arms: Sham tVNS

SUMMARY:
To verify the efficacy of transcutaneous vagus nerve stimulation (tVNS) on and autonomic balance in patients with chronic heart failure and reduced (HFrEF) or mildly reduced (HFmrEF) left ventricular ejection fraction. The study hypothesis is that tVNS increases baroreflex gain, with consequent benefits on sympathovagal balance (at short- and mid-term), and on quality of life and bio-humoral parameters (at mid-term).

DETAILED DESCRIPTION:
Pilot phase: comparing the effects of right- (10-minute) vs. left-sided tVNS (10-minute) on BRS and heart rate variability (HRV) in a subset of patients.

Short-term phase: comparing the effects of active- (10-minute) vs. sham-tVNS (10-minute) on BRS, HRV, and sympathetic nerve activity.

Mid-term phase: comparing the effects of active- (4-week) vs- sham-tVNS (4-week) on BRS, HRV, biomarkers, exercise performance, and cardiac function.

ELIGIBILITY:
Inclusion criteria

* Aged ≥18 years;
* Ability to consent to enrollment;
* Diagnosis of chronic heart failure (CHF= and left ventricular ejection fraction <50% according to the latest European guidelines.

Exclusion criteria

* History of acute coronary syndrome within 3 months of enrollment;
* Clinical need to modify CHF therapy during the study;
* History of recurrent syncope, orthostatic hypotension, severe bradycardia (average heart rate <50 bpm), or second or third-degree atrioventricular block;
* Neurological conditions characterized by dysautonomia (e.g., Parkinson's disease);
* Unstable major psychiatric disorders or treatment with psychoactive drugs or drugs that can act on the autonomic nervous system (e.g., antidepressants, antipsychotics, opioids, benzodiazepines);
* Uncontrolled thyroid disorders;
* Active neoplasia;
* Severe renal insufficiency (estimated glomerular filtration rate <15 ml/min/1.73 m2);
* Moderate or severe chronic obstructive pulmonary disease (FEV1/FVC <70% of predicted and FEV1 <70%);
* Liver insufficiency (AST/ALT >100 U/L and/or gamma-GT >150 U/L);
* Participation in other clinical studies in the 3 months preceding;
* Women in pregnancy, breastfeeding, or of childbearing age not following adequate contraception (the woman must agree to abstain from heterosexual intercourse or use at least two effective contraceptive measures such as bilateral tubal ligation, male sterilization, use of hormonal contraceptives that inhibit ovulation, intrauterine devices releasing hormones, copper intrauterine devices; all barrier devices must be used in combination with a spermicidal cream).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in baroreflex gain (ms/mmHg) | 10 minutes (short-term effect)
  Barorefex gain will be calculated calculated as the ratio between the standard deviation of RR intervals (ms) and systolic blood pressure (mmHg)
Mean change in baroreflex gain (ms/mmHg) | 4 weeks (mid-term effect)
  Barorefex gain will be calculated calculated as the ratio between the standard deviation of RR intervals (ms) and systolic blood pressure (mmHg)

OTHER OUTCOMES:
Mean change in MSNA burst incidence (bursts/100 heartbeats) | 10 minutes (short-term effect)
  Assessed through peroneal nerve microneurography (as previously detailed in doi: 10.3389/fphys.2022.934372).
Mean change in peak O2 consumption (mL/Kg/min) | 4 weeks (mid-term effect)
  Assessed through cardiopulmonary exercise test

CONTACTS AND LOCATIONS:
Locations (1):
- Michele Emdin, Pisa, Pi, Italy

IPD SHARING:
Plan to Share IPD: No